CLINICAL TRIAL: NCT02521870
Title: A Phase 1b/2, Open-label, Multicenter, Dose-escalation and Expansion Trial of Intratumoral SD-101 in Combination With Pembrolizumab in Patients With Metastatic Melanoma or Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (SYNERGY-001)
Brief Title: A Trial of Intratumoral Injections of SD-101 in Combination With Pembrolizumab in Patients With Metastatic Melanoma or Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A strategic restructuring including the planned conclusion of clinical oncology development programs and no further sponsoring of the development of SD-101.
Sponsor: Dynavax Technologies Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DV3-MEL-01; Keynote 184 (Other: Merck); SYNERGY-001 (Other: Dynavax)
Record Dates: First submitted 2015-07-30; First posted 2015-08-13 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Melanoma; Head Neck Cancer
Keywords: Skin Cancer; Skin Tumors; Head and Neck Squamous Cell Carcinoma; Cancer Immunotherapy
MeSH Terms: conditions — Melanoma; Head and Neck Neoplasms; Skin Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Dose Escalation Phase 1b (Experimental): Determine the maximum tolerated dose (MTD) of escalating doses of SD-101(1) administered in combination with pembrolizumab in patients with melanoma (anti-PD-1/L1 therapy naïve and experienced patients with progressive disease).
  Interventions: Drug: SD-101(1); Biological: Pembrolizumab
- Dose Expansion Phase 2 (Cohort 1) (Experimental): Determine the safety and efficacy of SD-101(2) and pembrolizumab in anti-PD-1/L1 therapy naïve patients with recurrent or metastatic melanoma.
  Interventions: Drug: SD-101(2); Biological: Pembrolizumab
- Dose Expansion Phase 2 (Cohort 2) (Experimental): Determine the safety and efficacy of SD-101(2) and pembrolizumab in anti-PD-1/L1 therapy progressing patients with recurrent or metastatic melanoma.
  Interventions: Drug: SD-101(2); Biological: Pembrolizumab
- Dose Expansion Phase 2 (Cohort 3) (Experimental): Determine the safety and efficacy of SD-101(2) and pembrolizumab in anti-PD-1/L1 therapy naïve patients with recurrent head and neck squamous cell carcinoma.
  Interventions: Drug: SD-101(2); Biological: Pembrolizumab
- Dose Expansion Phase 2 (Cohort 4) (Experimental): Determine the safety and efficacy of SD-101(2) and pembrolizumab in anti-PD-1/L1 therapy progressing patients with recurrent head and neck squamous cell carcinoma.
  Interventions: Drug: SD-101(2); Biological: Pembrolizumab
- Dose Expansion Phase 2 (Cohort 5) (Experimental): Determine the safety and efficacy of SD-101(3) and pembrolizumab in anti-PD-1/L1 therapy naïve patients with recurrent or metastatic melanoma.
  Interventions: Biological: SD-101(3); Biological: Pembrolizumab
- Dose Expansion Phase 2 (Cohort 6) (Experimental): Determine the safety and efficacy of SD-101(3) and pembrolizumab in anti-PD-1/L1 therapy naïve patients with recurrent head and neck squamous cell carcinoma.
  Interventions: Biological: SD-101(3); Biological: Pembrolizumab
- Dose Expansion Phase 2 (Cohort 7) (Experimental): Determine the safety and efficacy of SD-101(3) and pembrolizumab in anti-PD-1/L1 therapy refractory or resistant patients with recurrent head and neck squamous cell carcinoma.
  Interventions: Biological: SD-101(3); Biological: Pembrolizumab
- Dose Expansion Phase 2 (Cohort 8) (Experimental): Determine the safety and efficacy of SD-101(3) and pembrolizumab in anti-PD-1/L1 therapy refractory or resistant patients with recurrent or metastatic melanoma.
  Interventions: Biological: SD-101(3); Biological: Pembrolizumab

INTERVENTIONS:
Drug: SD-101(1) — SD-101 administered intratumorally at escalating doses (up to 11 doses).
  Arms: Dose Escalation Phase 1b
Biological: Pembrolizumab — Pembrolizumab administered intravenously, 200 mg Q3W for two years (up to 35 doses).
  Arms: Dose Escalation Phase 1b
Drug: SD-101(2) — Dose Q1W for 4 weeks followed by dose Q3W for 7 weeks, then 9 weeks off, then dose Q1W for 4 weeks followed by dose Q3W for 7 weeks (up to 22 total doses).
  Arms: Dose Expansion Phase 2 (Cohort 1); Dose Expansion Phase 2 (Cohort 2); Dose Expansion Phase 2 (Cohort 3); Dose Expansion Phase 2 (Cohort 4)
Biological: Pembrolizumab — Pembrolizumab administered intravenously, 200mg Q3W for two years (up to 35 doses).
  Arms: Dose Expansion Phase 2 (Cohort 1); Dose Expansion Phase 2 (Cohort 2); Dose Expansion Phase 2 (Cohort 3); Dose Expansion Phase 2 (Cohort 4)
Biological: SD-101(3) — Dose Q1W for 4 weeks followed by dose Q3W for 16 additional weeks (up to 20 total doses).
  Arms: Dose Expansion Phase 2 (Cohort 5); Dose Expansion Phase 2 (Cohort 6); Dose Expansion Phase 2 (Cohort 7); Dose Expansion Phase 2 (Cohort 8)
Biological: Pembrolizumab — Pembrolizumab administered intravenously, 200mg Q3W for two years (up to 35 doses).
  Arms: Dose Expansion Phase 2 (Cohort 5); Dose Expansion Phase 2 (Cohort 6); Dose Expansion Phase 2 (Cohort 7); Dose Expansion Phase 2 (Cohort 8)

SUMMARY:
This is a phase 1b/2, open-label, multicenter trial designed to evaluate the safety, tolerability, biologic activity, and preliminary efficacy of intratumoral SD-101 injections in combination with intravenous pembrolizumab in patients with metastatic melanoma or recurrent or metastatic head and neck squamous cell carcinoma (HNSCC).

This study will be conducted in 2 phases. Phase 1 evaluates SD-101 given in combination with pembrolizumab in melanoma populations (anti-PD-1/L1 naïve and anti-PD-1/L1 experienced with progressive disease) in up to 4 Dose Escalation cohorts to identify a recommended Phase 2 dose (RP2D) to be evaluated in up to 4 Dose Expansion cohorts in Phase 2. Phase 2 also includes up to 4 Dose Expansion cohorts of patients with HNSCC (anti-PD-1/L1 naïve and anti-PD-1/L1 experienced with progressive disease).

ELIGIBILITY:
[Inclusion Criteria (Phase 1 and Phase 2)]

1. Willing and able to provide written informed consent for the trial
2. Aged 18 years and older
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
4. Patient must have adequate organ function as indicated by the following laboratory values:

   1. Hematological:

      * Absolute neutrophil count (ANC) ≥ 1,500 /mcL
      * Platelet count ≥ 100,000 /mcL
      * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
   2. Renal:

      * Serum creatinine ≤ 1.5 × upper limit of normal (ULN) OR
      * Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥ 60 mL/min for subject with creatinine levels > 1.5 × institutional ULN
   3. Hepatic:

      * Serum total bilirubin:
      * ≤ 1.5 × ULN OR
      * < 3 × ULN for persons with Gilbert's syndrome OR
      * Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 × ULN
      * Aspartate transaminase (AST) and alanine transaminase (ALT) (also known as serum glutamic oxaloacetic transaminase and serum glutamic pyruvic transaminase)
      * ≤ 2.5 × ULN OR
      * ≤ 5 × ULN for patients with liver metastases
   4. Coagulation:

      * International normalized ratio or prothrombin time (PT) ≤ 1.5 × ULN unless patient is receiving anticoagulant therapy, and as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
      * Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless patient is receiving anticoagulant therapy, and as long as PT or PTT is within therapeutic range of intended use of anticoagulants
5. Have provided 2 tissue biopsy samples taken of the target lesion (Lesion A) as a single biopsy split into 2 samples or 2 separate biopsies that meet the minimal sample size requirement per the study laboratory manual. One sample is for determining PD-L1 expression level by immunohistochemistry and can be an archival sample of the anticipated target lesion that has been collected within 3 months of screening. The other sample is for RNA expression profiling and must be a fresh biopsy.
6. Life expectancy of at least 6 months
7. Female patients of childbearing potential, as defined in Section 5.2.1, must have a negative urine or serum pregnancy test within 72 hours prior to taking the first dose of trial treatment. If the urine test is positive or cannot be confirmed as negative then a serum test is required which must be negative for the patient to enroll. Women of childbearing potential (WOCBP) must be willing to use 2 medically acceptable methods of contraceptive from Day 1 through 120 days after the last dose of trial treatment. The 2 medically acceptable birth control methods can be either 2 barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide as per local regulations or guidelines. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).

   Male patients of reproductive potential, as described in Section 5.2.1, must agree to use an adequate method of contraception from Day 1 through 120 days after the last dose of trial treatment.

   Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

   [Inclusion Criteria (Phase 1 only: Melanoma)]
8. Histologically or cytologically confirmed unresectable or metastatic (stage IV) melanoma
9. For Phase 1 Escalation Cohorts 1-4, must have at least 1 lesion that qualifies as a target lesion per RECIST v1.1 except for the minimum measurement of 10 mm in diameter for superficial lesions, is easily accessible (palpable or can be visualized by ultrasound), and is amenable to multiple intratumoral injections. If superficial, the target lesion must be documented photographically.

   [Inclusion Criteria (Phase 2 only: Melanoma)]
10. Histologically or cytologically confirmed recurrent or unresectable or metastatic (stage IV) melanoma
11. Must have at least 2 lesions that qualify as a target lesion per RECIST v1.1, and 1 of the qualifying lesions must be easily accessible (palpable or can be visualized by ultrasound) and amenable to multiple intratumoral injections. The target lesion should be of sufficient size such that the required tumor biopsies do not significantly affect tumor assessment per RECIST v1.1. If superficial, the target lesion must measure at least 10 mm in diameter, be measured by calipers, and be documented photographically. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion. Approval from the Medical Monitor is required to inject a previously radiated lesion.
12. Expansion Cohort 2: Must have documented PD per RECIST v1.1 on a prior treatment regimen containing an anti-PD-1/L1 drug (see Appendix 6 for definition of PD per RECIST v1.1)
13. Expansion Cohort 8: Must have all of the following:

    1. Received at least 2 doses of an anti-PD-1/L1 therapy
    2. PD occurred within 3 months after last dose of anti-PD-1/L1 therapy
    3. Documented PD per RECIST v.1.1, which has been confirmed by a second assessment at least 4 weeks from the date of the first documented PD, in the absence of rapid clinical progression

    [Inclusion Criteria (Phase 2 only: HNSCC)]
14. Histologically or cytologically confirmed recurrent or metastatic HNSCC that could not be treated with curative intent
15. Must have at least 1 lesion that qualifies as a target lesion per RECIST v1.1, and which must be easily accessible (palpable or can be visualized by ultrasound) and amenable to multiple intratumoral injections. The target lesion should be of sufficient size such that the required tumor biopsies do not significantly affect tumor assessment per RECIST v1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion. Approval from the Medical Monitor is required to inject a previously radiated lesion.
16. Expansion Cohort 4: Must have documented confirmed PD per RECIST v1.1 on a prior treatment regimen containing an anti-PD-1/L1 drug (see Appendix 6 for definition of PD per RECIST v1.1)
17. Expansion Cohort 7: Must have all of the following:

    1. Received at least 2 doses of an anti-PD-1/L1 therapy, where the last dose of anti-PD-1/L1 therapy was within 6 months of study enrollment (Day 1)
    2. Refractory response, ie, PD occurred within 3 months duration of the start of treatment on anti-PD-1/L1 therapy; OR resistant response, ie, PD occurred beyond 3 months duration of treatment on anti-PD-1/L1 therapy and within 6 months after the last dose of treatment on anti-PD-1/L1 therapy
    3. Documented PD per RECIST v.1.1, which has been confirmed by a second assessment at least 4 weeks from the date of the first documented PD, in the absence of rapid clinical progression

[Exclusion Criteria (Phase 1 and Phase 2)]

1. Received systemic chemotherapy or biological cancer therapy (except anti-PD-1/L1 therapy) within 3 weeks prior to study enrollment
2. Received prior radiotherapy within 2 weeks of start of study therapy. A shorter washout period may be permitted after approval by the Medical Monitor.
3. Received small molecule inhibitor targeted therapy, such as tyrosine kinase inhibitors, within 2 weeks prior to study enrollment
4. Has not recovered to CTCAE Grade 1 or better from the AEs due to cancer therapeutics prior to study enrollment

   NOTE: Patients with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia or Grade 2 AEs that qualify as Grade 2 due to replacement hormonal or steroid therapy are exceptions to this criterion and may qualify for the study with approval by a Dynavax Medical Monitor.

   If a patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to enrollment.
5. Received a transfusion of blood products (including platelets or red blood cells) or colony-stimulating factors (including G-CSF, GM-CSF or recombinant erythropoietin) within 4 weeks prior to study enrollment
6. Is expected to require any other form of anti-cancer therapy while in the trial
7. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy (including immune modulators or systemic corticosteroids) within 7 days prior to study enrollment
8. Positive for active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection as determined by laboratory tests for HBsAg, anti-HBc, and anti-HBs; anti-HCV; and anti-HIV -1/2, respectively
9. History of or current uveal or ocular or mucosal melanoma
10. Active infection including cytomegalovirus
11. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial through 120 days after the last dose of trial treatment
12. Active autoimmune disease requiring systemic treatment in the past 2 years or a disease that requires immunosuppressive medication including systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
13. Current pneumonitis or history of (non-infectious) pneumonitis that required steroids
14. An immune-related AE from a previous immunotherapeutic agent that has not resolved to Grade 1 or less prior to study enrollment. The exception is a Grade 2 AE which qualifies as Grade 2 due to replacement steroid therapy which may be allowed with approval by a Dynavax Medical Monitor.
15. Known active central nervous system metastases or carcinomatous meningitis

    NOTE: Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging [using the identical imaging modality for each assessment, either MRI or CT scan] for at least 4 weeks prior to the first dose of trial treatment and with any neurologic symptoms returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
16. Use of any investigational agent within the last 28 days prior to study enrollment
17. Has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
18. Any other significant medical or psychiatric condition, laboratory abnormality, or difficulty complying with protocol requirements that may increase the risk associated with trial participation or trial drug administration that may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for this trial
19. History of sensitivity to any component of SD-101 or hypersensitivity reaction to treatment with a monoclonal antibody and/or any of its excipients
20. Any known additional malignancy that is progressing or requires active treatment. Exceptions are cutaneous melanoma or HNSCC under study per protocol, or basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ cervical cancer that has undergone potentially curative therapy.

    [Exclusion Criteria (Phase 2, Melanoma Expansion Cohorts 1 and 5 only)]
21. Melanoma considered resectable with curative intent
22. Prior therapy with an anti-PD-1/L1 agent
23. Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients

    [Exclusion Criteria (Phase 2, Melanoma Expansion Cohorts 2 and 8 only)]
24. Melanoma considered resectable with curative intent
25. Any prior combination therapy involving agents given by intratumoral injection that target the innate immune pathway or system such as oncolytic viral or microbial therapy (eg, T-VEC [talimogene laherparepvec]), toll-like receptors (TLR) agonists, STING or RIG-1 and an anti-PD-1/L1 inhibitor

    [Exclusion Criteria (Phase 2, HNSCC Expansion Cohorts 3 and 6 only)]
26. HNSCC considered resectable with curative intent
27. Prior therapy with an anti-PD-1/L1 agent
28. Require anticoagulation therapy

    [Exclusion Criteria (Phase 2, HNSCC Expansion Cohorts 4 and 7 only)]
29. HNSCC considered resectable with curative intent
30. Any prior combination therapy involving agents given by intratumoral injection that target the innate immune pathway or system such as oncolytic viral or microbial therapy (eg, T-VEC), TLR agonists, STING or RIG-1 and an anti-PD-1/L1 inhibitor
31. Require treatment on anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2015-09; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, MD, Principal Investigator — UCLA School of Medicine (Melanoma); Ezra Cohen, MD, Principal Investigator — UCSD Moores Cancer Center (HNSCC); Thomas Tüting, MD, Principal Investigator — University Hospital Magdeburg
Locations (47):
- United States (30):
  - University of Alabama School of Medicine, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - Stanford Hospitals and Clinics, Palo Alto, California
  - University of California, San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Georgia Cancer Center - Northside Hospital Central Research Department, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa Healthcare, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Atlantic Health, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center - Seidman Cancer center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - University of Utah Health Care - Huntsman Cancer institute, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - West Virginia University, Morgantown, West Virginia
- Australia (5):
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Liverpool Hospital, Westmead, New South Wales
  - Melanoma Institute, Wollstonecraft, New South Wales
  - Adelaide Cancer Centre - Ashford Cancer Centre, Kurralta Park, South Australia
  - Hollywood Private Hospital / Affinity Research, Nedlands, Western Australia
- Germany (9):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum BuxtehudeDermato-Onkologie Studienzentrale, Buxtehude
  - Uniklinikum Dresden Klinik und Poliklinik für Dermatologie, Dresden
  - Universitätshautklinik Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - HNO-Universitätsklinik Jena, Jena
  - Universitätshautklinik Magdeburg, Magdeburg
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared under guidance of the New Rule - FDAAA 801 eff. Jan 2017. 3/2017 - additional changes forthcoming.

REFERENCES:
- [Derived] Ribas A, Medina T, Kummar S, Amin A, Kalbasi A, Drabick JJ, Barve M, Daniels GA, Wong DJ, Schmidt EV, Candia AF, Coffman RL, Leung ACF, Janssen RS. SD-101 in Combination with Pembrolizumab in Advanced Melanoma: Results of a Phase Ib, Multicenter Study. Cancer Discov. 2018 Oct;8(10):1250-1257. doi: 10.1158/2159-8290.CD-18-0280. Epub 2018 Aug 28. PMID 30154193

RESULTS

PARTICIPANT FLOW:
Groups:
- SD-101 1 mg: Dose Escalation Cohort 4: Participants were administered SD-101 1 mg intratumorally as 4 weekly doses followed by 1 dose Q3W for 7 additional doses. Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 2 mg: Dose Escalation Cohort 1: Participants were administered SD-101 2 mg intratumorally as 4 weekly doses followed by 1 dose Q3W for 7 additional doses. Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 4 mg: Dose Escalation Cohort 2: Participants were administered SD-101 4 mg intratumorally as 4 weekly doses followed by 1 dose Q3W for 7 additional doses. Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 8 mg: Dose Escalation Cohort 3: Participants were administered SD-101 8 mg intratumorally as 4 weekly doses followed by 1 dose Q3W for 7 additional doses. Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 8 mg in Anti-PD-1/L1-Naïve Melanoma: Dose Expansion Cohort 1: Participants with melanoma who are anti-PD-1/L1-naïve were administered SD-101 8 mg intratumorally starting on Day 22 dose Q1W for 4 weeks followed by dose Q3W for 7 doses, then 9 weeks off, then dose Q1W for 4 weeks followed by dose Q3W for 7 doses (up to 22 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 8 mg in Anti-PD-1/L1-Experienced Melanoma: Dose Expansion Cohort 2: Participants with melanoma who are anti-PD-1/L1-experienced were administered SD-101 8 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 7 doses, then 9 weeks off, then dose Q1W for 4 weeks followed by dose Q3W for 7 doses (up to 22 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 8 mg in Anti-PD-1/L1-Naïve HNSCC: Dose Expansion Cohort 3: Participants with HNSCC who are anti-PD-1/L1-naïve were administered SD-101 8 mg intratumorally starting on Day 22 dose Q1W for 4 weeks followed by dose Q3W for 7 doses, then 9 weeks off, then dose Q1W for 4 weeks followed by dose Q3W for 7 doses (up to 22 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 8 mg in Anti-PD-1/L1-Experienced HNSCC: Dose Expansion Cohort 4: Participants with HNSCC who are anti-PD-1/L1-experienced were administered SD-101 8 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 7 doses, then 9 weeks off, then dose Q1W for 4 weeks followed by dose Q3W for 7 doses (up to 22 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 2 mg in Anti-PD-1/L1-Naïve Melanoma: Dose Expansion Cohort 5: Participants with melanoma who are anti-PD-1/L1-naïve were administered SD-101 2 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 16 doses (up to 20 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 2 mg in Anti-PD-1/L1-Naïve HNSCC: Dose Expansion Cohort 6: Participants with HNSCC who are anti-PD-1/L1-naïve were administered SD-101 2 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 16 doses (up to 20 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant HNSCC: Dose Expansion Cohort 7: Participants with HNSCC who are anti-PD-1/L1 refractory or resistant were administered SD-101 2 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 16 doses (up to 20 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant Melanoma: Dose Expansion Cohort 8: Participants with melanoma who are anti-PD-1/L1 refractory or resistant were administered SD-101 2 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 16 doses (up to 20 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
Period: Phase 1: Dose Escalation
Arm/Group | SD-101 1 mg | SD-101 2 mg | SD-101 4 mg | SD-101 8 mg | SD-101 8 mg in Anti-PD-1/L1-Naïve Melanoma | SD-101 8 mg in Anti-PD-1/L1-Experienced Melanoma | SD-101 8 mg in Anti-PD-1/L1-Naïve HNSCC | SD-101 8 mg in Anti-PD-1/L1-Experienced HNSCC | SD-101 2 mg in Anti-PD-1/L1-Naïve Melanoma | SD-101 2 mg in Anti-PD-1/L1-Naïve HNSCC | SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant HNSCC | SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant Melanoma
Started | 6 | 5 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed SD-101 Treatment (up to 11 Doses) | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed Pembrolizumab Treatment (up to 35 doses)) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 4 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 2 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2: Dose Expansion
Arm/Group | SD-101 1 mg | SD-101 2 mg | SD-101 4 mg | SD-101 8 mg | SD-101 8 mg in Anti-PD-1/L1-Naïve Melanoma | SD-101 8 mg in Anti-PD-1/L1-Experienced Melanoma | SD-101 8 mg in Anti-PD-1/L1-Naïve HNSCC | SD-101 8 mg in Anti-PD-1/L1-Experienced HNSCC | SD-101 2 mg in Anti-PD-1/L1-Naïve Melanoma | SD-101 2 mg in Anti-PD-1/L1-Naïve HNSCC | SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant HNSCC | SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant Melanoma
Started | 0 | 0 | 0 | 0 | 57 | 25 | 23 | 9 | 24 | 28 | 23 | 30
Completed SD-101 Treatment (up to 11 Doses) | 0 | 0 | 0 | 0 | 25 | 7 | 3 | 2 | 9 | 5 | 1 | 11
Completed SD-101 Treatment Cycle 2 (up to 22 Doses) | 0 | 0 | 0 | 0 | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed Pembrolizumab Treatment (up to 35 doses)) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 2 (4 participants completed pembrolizumab treatment (up to 35 cycles).) | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 52 | 25 | 23 | 9 | 22 | 28 | 23 | 30
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 0 | 1 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 11 | 2 | 0 | 1 | 5 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 22 | 18 | 17 | 7 | 5 | 17 | 17 | 21
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 5 | 2 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 10 | 3 | 2 | 0 | 10 | 5 | 1 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population comprises all participants who received at least one dose of SD-101. Phase 1 Dose Escalation cohorts and Phase 2 Dose Expansion cohorts were rearranged as analysis groups for analyses to assess study objectives, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101, as specified by the statistical analysis plan. Participants who received 1 mg or 4 mg of SD-101 in Phase 1: Dose Escalation of the study are not included in the analysis groups.
Groups:
- Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg: Phase 1 Dose Escalation cohorts and Phase 2 Dose Expansion cohorts were rearranged as analysis groups for analyses to assess study objectives, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101.
  The participants in this analysis group include participants in Phase 1 Dose Escalation Cohort 1 (SD-101 2 mg) and participants in Phase 2 Dose Expansion Cohort 1 and Cohort 5.
- Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg: Phase 1 Dose Escalation cohorts and Phase 2 Dose Expansion cohorts were rearranged as analysis groups for analyses to assess study objectives, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101.
  The participants in this analysis group include participants in Phase 1 Dose Escalation Cohort 3 (SD-101 8 mg) and participants in Phase 2 Dose Expansion Cohort 1.
- Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg: Phase 1 Dose Escalation cohorts and Phase 2 Dose Expansion cohorts were rearranged as analysis groups for analyses to assess study objectives, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101.
  The participants in this analysis group include participants in Phase 1 Dose Escalation Cohort 1 (SD-101 2 mg) and participants in Phase 2 Dose Expansion Cohort 2 and Cohort 8.
- Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg: Phase 1 Dose Escalation cohorts and Phase 2 Dose Expansion cohorts were rearranged as analysis groups for analyses to assess study objectives, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101.
  The participants in this analysis group include participants in Phase 1 Dose Escalation Cohort 3 (SD-101 8 mg) and participants in Phase 2 Dose Expansion Cohort 2.
- HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg: Phase 1 Dose Escalation cohorts and Phase 2 Dose Expansion cohorts were rearranged as analysis groups for analyses to assess study objectives, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101.
  The participants in this analysis group include participants in Phase 2 Dose Expansion Cohort 3 and Cohort 6.
- HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg: Phase 1 Dose Escalation cohorts and Phase 2 Dose Expansion cohorts were rearranged as analysis groups for analyses to assess study objectives, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101.
  The participants in this analysis group include participants in Phase 2 Dose Expansion Cohort 3.
- HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg: Phase 1 Dose Escalation cohorts and Phase 2 Dose Expansion cohorts were rearranged as analysis groups for analyses to assess study objectives, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101.
  The participants in this analysis group include participants in Phase 2 Dose Expansion Cohort 4 and Cohort 7.
- HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg: Phase 1 Dose Escalation cohorts and Phase 2 Dose Expansion cohorts were rearranged as analysis groups for analyses to assess study objectives, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101.
  The participants in this analysis group include participants in Phase 2 Dose Expansion Cohort 4.
- Total: Total of all reporting groups
Arm/Group | Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg | Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg | Total
Number analyzed (Participants) | 45 | 41 | 31 | 30 | 28 | 23 | 23 | 9 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 13 | 17 | 16 | 10 | 15 | 4 | 109
  >=65 years | 29 | 23 | 18 | 13 | 12 | 13 | 8 | 5 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (13.34) | 65.3 (12.44) | 65.6 (12.99) | 62.4 (15.25) | 62.6 (10.66) | 67.2 (9.59) | 61.0 (12.94) | 65.2 (12.35) | 64.4 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 10 | 7 | 9 | 2 | 8 | 1 | 64
  Male | 32 | 27 | 21 | 23 | 19 | 21 | 15 | 8 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 4 | 0 | 0 | 2 | 1 | 10
  Not Hispanic or Latino | 43 | 37 | 28 | 26 | 28 | 22 | 20 | 8 | 212
  Unknown or Not Reported | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 41 | 30 | 25 | 24 | 20 | 19 | 9 | 212
  Black or African American | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 5
  Asian | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 7
  Other | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 6
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG PS = Eastern Cooperative Oncology Group Performance Status; 0 = Fully active, able to carry on all pre-disease performance without restriction (better outcome)
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work (worse outcome)
  Participants
    0 | 28 | 30 | 19 | 16 | 5 | 6 | 4 | 2 | 110
    1 | 17 | 11 | 12 | 14 | 23 | 17 | 19 | 7 | 120
PDL1 Expression [Count of Participants; unit: Participants]
  Positive | 21 | 13 | 9 | 13 | 14 | 15 | 4 | 7 | 96
  Negative | 14 | 15 | 8 | 11 | 2 | 4 | 5 | 1 | 60
  Unknown | 10 | 13 | 14 | 6 | 12 | 4 | 14 | 1 | 74

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Dose Escalation Only - Number of Participants With DLTs
Description: Dose-limiting toxicities (DLTs) are defined per protocol as specific AEs occurring from the time of the first injection (Day 1) through Day 29.
Time Frame: Day 1 through Day 29
Population: The safety population is defined as comprising of participants who received at least 1 dose of SD-101.
Measure: Count of Participants; unit: Participants
Groups:
- SD-101 8 mg in Anti-PD-1/L1-Naïve Melanoma: Dose Expansion Cohort 1: Participants with melanoma who are anti-PD-1/L1-naïve were administered SD-101 8 mg intratumorally starting on Day 22 dose Q1W for 4 weeks followed by dose Q3W for 7 weeks, then 9 weeks off, then dose Q1W for 4 weeks followed by dose Q3W for 7 weeks (up to 22 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 8 mg in Anti-PD-1/L1-Experienced Melanoma: Dose Expansion Cohort 2: Participants with melanoma who are anti-PD-1/L1-experienced were administered SD-101 8 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 7 weeks, then 9 weeks off, then dose Q1W for 4 weeks followed by dose Q3W for 7 weeks (up to 22 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 8 mg in Anti-PD-1/L1-Naïve HNSCC: Dose Expansion Cohort 3: Participants with HNSCC who are anti-PD-1/L1-naïve were administered SD-101 8 mg intratumorally starting on Day 22 dose Q1W for 4 weeks followed by dose Q3W for 7 weeks, then 9 weeks off, then dose Q1W for 4 weeks followed by dose Q3W for 7 weeks (up to 22 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 8 mg in Anti-PD-1/L1-Experienced HNSCC: Dose Expansion Cohort 4: Participants with HNSCC who are anti-PD-1/L1-experienced were administered SD-101 8 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 7 weeks, then 9 weeks off, then dose Q1W for 4 weeks followed by dose Q3W for 7 weeks (up to 22 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 2 mg in Anti-PD-1/L1-Naïve Melanoma: Dose Expansion Cohort 5: Participants with melanoma who are anti-PD-1/L1-naïve were administered SD-101 2 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 16 weeks (up to 20 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 2 mg in Anti-PD-1/L1-Naïve HNSCC: Dose Expansion Cohort 6: Participants with HNSCC who are anti-PD-1/L1-naïve were administered SD-101 2 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 16 weeks (up to 20 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant HNSCC: Dose Expansion Cohort 7: Participants with HNSCC who are anti-PD-1/L1 refractory or resistant were administered SD-101 2 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 16 weeks (up to 20 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
- SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant Melanoma: Dose Expansion Cohort 8: Participants with melanoma who are anti-PD-1/L1 refractory or resistant were administered SD-101 2 mg intratumorally starting on Day 1 dose Q1W for 4 weeks followed by dose Q3W for 16 weeks (up to 20 total doses). Participants were also administered Pembrolizumab 200 mg intravenously Q3W starting on Day 1 for up to 35 treatments or until disease progression.
Arm/Group | SD-101 1 mg | SD-101 2 mg | SD-101 4 mg | SD-101 8 mg | SD-101 8 mg in Anti-PD-1/L1-Naïve Melanoma | SD-101 8 mg in Anti-PD-1/L1-Experienced Melanoma | SD-101 8 mg in Anti-PD-1/L1-Naïve HNSCC | SD-101 8 mg in Anti-PD-1/L1-Experienced HNSCC | SD-101 2 mg in Anti-PD-1/L1-Naïve Melanoma | SD-101 2 mg in Anti-PD-1/L1-Naïve HNSCC | SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant HNSCC | SD-101 2 mg in Anti-PD-1/L1 Refractory or Resistant Melanoma
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1 Dose Escalation and Phase 2 Dose Expansion - Overall Response Rate (ORR) by Analysis Group
Description: Overall response rate (ORR) by analysis group based on investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 was evaluated from Baseline (Day 1) through Day 743 or End of Study (EOS).
Time Frame: Day 1 through Day 743
Population: The intent-to-treat (ITT) population comprises of all participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg | Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg
Number analyzed (Participants) | 45 | 41 | 31 | 30 | 28 | 23 | 23 | 9
Participants
  Complete Response | 9 | 4 | 0 | 1 | 2 | 0 | 0 | 1
  Partial Response | 25 | 16 | 7 | 3 | 4 | 6 | 2 | 0
  Stable Disease | 2 | 8 | 8 | 8 | 7 | 5 | 3 | 2
  Progressive Disease | 5 | 8 | 12 | 11 | 10 | 9 | 10 | 4
  Not Evaluable | 4 | 5 | 4 | 7 | 5 | 3 | 8 | 2

3. Secondary Outcome: Phase 1 Dose Escalation and Phase 2 Dose Expansion - Time to Objective Response by Analysis Group
Description: Time to objective response by analysis group based on investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 was evaluated from Baseline (Day 1) through Day 743 or End of Study (EOS).
Time Frame: Day 1 through Day 743
Population: The intent-to-treat (ITT) population comprises of all participants who were enrolled in the study. This subset of participants analyzed comprises of participants with objective response.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg | Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg
Number analyzed (Participants) | 34 | 20 | 7 | 4 | 6 | 6 | 2 | 1
months | 3.2 (1.6) | 4.1 (2.96) | 5.1 (3.06) | 4.3 (2.98) | 2.3 (.92) | 2.4 (0.87) | 2.7 (1.09) | 2.1 (0)

4. Secondary Outcome: Phase 1 Dose Escalation and Phase 2 Dose Expansion - Duration of Response by Analysis Group
Description: Duration of response by analysis group based on investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 was evaluated from Baseline (Day 1) through Day 743 or End of Study (EOS).
Time Frame: Day 1 through Day 743
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg | Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg
Number analyzed (Participants) | 34 | 20 | 7 | 4 | 6 | 6 | 2 | 1
months | 11.1 (6.42) | 11.7 (5.96) | 4.6 (6.57) | 7.6 (7.28) | 5.9 (4.93) | 6.3 (3.96) | 2.1 (0.07) | 8.1 (0)

5. Secondary Outcome: Phase 1 Dose Escalation and Phase 2 Dose Expansion - Disease Control Rate (DCR) by Analysis Group
Description: Disease Control Rate (DCR) by analysis group based on investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 was evaluated from Baseline (Day 1) through Day 743 or End of Study (EOS).
Time Frame: Day 1 through Day 743
Population: The intent-to-treat (ITT) population comprises of all participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg | Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg
Number analyzed (Participants) | 45 | 41 | 31 | 30 | 28 | 23 | 23 | 9
Participants | 36 | 28 | 15 | 12 | 13 | 11 | 5 | 3

6. Secondary Outcome: Phase 1 Dose Escalation and Phase 2 Dose Expansion - Progression-Free Survival Rate by Analysis Group
Description: Progression-Free Survival (PFS) rate by analysis group based on investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 was evaluated from Baseline (Day 1) through Day 743 or End of Study (EOS).
Time Frame: Day 1 through Day 743
Population: The intent-to-treat (ITT) population comprises of all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg | Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg
Number analyzed (Participants) | 45 | 41 | 31 | 30 | 28 | 23 | 23 | 9
percentage of participants
  3 months | 85.7 [70.9 to 93.3] | 71.9 [54 to 83.8] | 46.7 [28.4 to 63] | 48 [27.8 to 65.6] | 46.4 [26.6 to 64.1] | 43.5 [23.3 to 62.1] | 31.6 [12.9 to 52.2] | 37.5 [8.7 to 67.4]
  6 months | 78.4 [62.6 to 88.1] | 63.3 [45.2 to 76.8] | 33 [17.2 to 49.8] | 24 [9.8 to 41.7] | 26.5 [10.5 to 45.7] | 17.4 [5.4 to 35] | 0 [0 to 0] | 25 [3.7 to 55.8]
  9 months | 70.8 [54.3 to 82.3] | 60.4 [42.4 to 74.4] | 21.4 [8.6 to 37.9] | 14.4 [3.9 to 31.4] | 21.2 [7.1 to 40.3] | 17.4 [5.4 to 35] | 0 [0 to 0] | 12.5 [0.7 to 42.3]
  12 months | 70.8 [54.3 to 82.3] | 53.7 [35.7 to 68.7] | 21.4 [8.6 to 37.9] | 9.6 [1.7 to 25.7] | 15.9 [4.2 to 34.4] | 8.7 [1.5 to 24.2] | 00 [0 to 0] | 0 [0 to 0]
  15 months | 65.1 [48.2 to 77.8] | 49.9 [31.9 to 65.5] | 0 [0 to 0] | 9.6 [1.7 to 25.7] | 15.9 [4.2 to 34.4] | 4.3 [0.3 to 18.2] | 00 [0 to 0] | 0 [0 to 0]
  18 months | 61.5 [44 to 75] | 40.3 [22.3 to 57.7] | 0 [0 to 0] | 9.6 [1.7 to 25.7] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  21 months | 61.5 [44 to 75] | 40.3 [22.3 to 57.7] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  24 months | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: From informed consent through Day 743
Groups:
- Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg: Some of the Phase 1 dose escalation cohorts and the 8 Phase 2 dose expansion cohorts were rearranged as analysis groups for analyses to assess the Phase 2 objectives as specified by the statistical analysis plan, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101. Results for Phase 2 objectives, using combined Phases 1 and 2 data, are presented by 2mg/lesion and 8mg/lesion doses.
  The participants in this analysis group include participants in Phase 1 Dose Escalation Cohort 1 (SD-101 2 mg) and participants in Phase 2 Dose Expansion Cohort 5.
- Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg: Some of the Phase 1 dose escalation cohorts and the 8 Phase 2 dose expansion cohorts were rearranged as analysis groups for analyses to assess the Phase 2 objectives as specified by the statistical analysis plan, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101. Results for Phase 2 objectives, using combined Phases 1 and 2 data, are presented by 2mg/lesion and 8mg/lesion doses.
  The participants in this analysis group include participants in Phase 1 Dose Escalation Cohort 3 (SD-101 8 mg) and participants in Phase 2 Dose Expansion Cohort 1.
- Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg: Some of the Phase 1 dose escalation cohorts and the 8 Phase 2 dose expansion cohorts were rearranged as analysis groups for analyses to assess the Phase 2 objectives as specified by the statistical analysis plan, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101. Results for Phase 2 objectives, using combined Phases 1 and 2 data, are presented by 2mg/lesion and 8mg/lesion doses.
  The participants in this analysis group include participants in Phase 1 Dose Escalation Cohort 1 (SD-101 2 mg) and participants in Phase 2 Dose Expansion Cohort 8.
- Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg: Some of the Phase 1 dose escalation cohorts and the 8 Phase 2 dose expansion cohorts were rearranged as analysis groups for analyses to assess the Phase 2 objectives as specified by the statistical analysis plan, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101. Results for Phase 2 objectives, using combined Phases 1 and 2 data, are presented by 2mg/lesion and 8mg/lesion doses.
  The participants in this analysis group include participants in Phase 1 Dose Escalation Cohort 3 (SD-101 8 mg) and participants in Phase 2 Dose Expansion Cohort 2.
- HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg: Some of the Phase 1 dose escalation cohorts and the 8 Phase 2 dose expansion cohorts were rearranged as analysis groups for analyses to assess the Phase 2 objectives as specified by the statistical analysis plan, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101. Results for Phase 2 objectives, using combined Phases 1 and 2 data, are presented by 2mg/lesion and 8mg/lesion doses.
  The participants in this analysis group include participants in Phase 2 Dose Expansion Cohort 6.
- HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg: Some of the Phase 1 dose escalation cohorts and the 8 Phase 2 dose expansion cohorts were rearranged as analysis groups for analyses to assess the Phase 2 objectives as specified by the statistical analysis plan, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101. Results for Phase 2 objectives, using combined Phases 1 and 2 data, are presented by 2mg/lesion and 8mg/lesion doses.
  The participants in this analysis group include participants in Phase 2 Dose Expansion Cohort 3.
- HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg: Some of the Phase 1 dose escalation cohorts and the 8 Phase 2 dose expansion cohorts were rearranged as analysis groups for analyses to assess the Phase 2 objectives as specified by the statistical analysis plan, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101. Results for Phase 2 objectives, using combined Phases 1 and 2 data, are presented by 2mg/lesion and 8mg/lesion doses.
  The participants in this analysis group include participants in Phase 2 Dose Expansion and Cohort 7.
- HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg: Some of the Phase 1 dose escalation cohorts and the 8 Phase 2 dose expansion cohorts were rearranged as analysis groups for analyses to assess the Phase 2 objectives as specified by the statistical analysis plan, based on tumor indications, anti-PD-1/L1 experience, and dose of SD-101. Results for Phase 2 objectives, using combined Phases 1 and 2 data, are presented by 2mg/lesion and 8mg/lesion doses.
  The participants in this analysis group include participants in Phase 2 Dose Expansion Cohort 4.
Arm/Group | Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg | Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg | Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg | HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg | HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg
All-Cause Mortality (participants affected / at risk) | 2/44 | 3/39 | 5/31 | 7/30 | 6/27 | 13/23 | 7/23 | 3/9
Serious Adverse Events (participants affected / at risk) | 15/44 | 17/39 | 6/31 | 9/30 | 8/27 | 5/23 | 10/23 | 4/9
Other Adverse Events (participants affected / at risk) | 44/44 | 39/39 | 31/31 | 30/30 | 25/27 | 23/23 | 22/23 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg (N=44) | Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg (N=39) | Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg (N=31) | Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg (N=30) | HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg (N=27) | HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg (N=23) | HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg (N=23) | HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Autoimmune myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune retinopathy (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 3 | 2 | 1 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Violence-related symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arterial rupture (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Melanoma Anti-PD-1/L1 Naïve SD-101 2 mg (N=44) | Melanoma Anti-PD-1/L1 Naïve SD-101 8 mg (N=39) | Melanoma Anti-PD-1/L1 Experienced SD-101 2 mg (N=31) | Melanoma Anti-PD-1/L1 Experienced SD-101 8 mg (N=30) | HNSCC Anti-PD-1/L1 Naïve SD-101 2 mg (N=27) | HNSCC Anti-PD-1/L1 Naïve SD-101 8 mg (N=23) | HNSCC Anti-PD-1/L1 Experienced SD-101 2 mg (N=23) | HNSCC Anti-PD-1/L1 Experienced SD-101 8 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 7 | 10 | 4 | 4 | 4 | 5 | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 11 | 3 | 1 | 1 | 2 | 2 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 2 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 3 | 2 | 6 | 4 | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 11 | 6 | 7 | 2 | 7 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 5 | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 15 | 9 | 10 | 8 | 8 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 6 | 6 | 6 | 5 | 3 | 0 | 0
Asthenia (General disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 19 | 20 | 6 | 16 | 3 | 10 | 2 | 1
Face oedema (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 33 | 31 | 13 | 22 | 15 | 17 | 7 | 5
Gait disturbance (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 13 | 7 | 10 | 4 | 2 | 2 | 0 | 0
Injection site erythema (General disorders) | 17 | 9 | 4 | 13 | 1 | 4 | 2 | 1
Injection site induration (General disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 11 | 6 | 4 | 8 | 0 | 0 | 2 | 1
Injection site pruritus (General disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 9 | 5 | 0 | 0 | 2 | 3 | 1 | 1
Malaise (General disorders) | 14 | 20 | 4 | 11 | 0 | 0 | 2 | 2
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 4 | 5 | 2 | 2 | 1 | 2 | 0 | 0
Pain (General disorders) | 5 | 3 | 2 | 2 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 10 | 15 | 7 | 7 | 6 | 6 | 6 | 4
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Candida infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 1 | 1 | 1 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 3 | 2 | 3 | 1 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2 | 1 | 2 | 2 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 5 | 2 | 4 | 2 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 7 | 8 | 0 | 0 | 1 | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 2 | 1 | 3 | 2 | 1 | 0 | 0
Platelet count decreased (Investigations) | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Tri-iodothyronine free decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 4 | 2 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 11 | 11 | 3 | 9 | 3 | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 4 | 0 | 0 | 1 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4 | 2 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 3 | 1 | 2 | 3 | 2 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 8 | 3 | 4 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 3 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 17 | 2 | 16 | 1 | 9 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1 | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 4 | 2 | 4 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 7 | 5 | 3 | 4 | 5 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 23 | 25 | 9 | 14 | 3 | 10 | 2 | 4
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Tremor (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2
Insomnia (Psychiatric disorders) | 4 | 4 | 3 | 1 | 3 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 3 | 6 | 3 | 2 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 6 | 4 | 0 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0 | 2 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 3 | 4 | 3 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 6 | 3 | 7 | 2 | 4 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 11 | 7 | 1 | 1 | 2 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 5 | 3 | 3 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 13 | 1 | 2 | 1 | 2 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 1
Lymphoedema (Vascular disorders) | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The sponsor terminated the trial early due to strategic restructuring, including the planned conclusion of clinical oncology development programs and no further sponsoring of the development of SD-101.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT02521870/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT02521870/SAP_001.pdf